CLINICAL TRIAL: NCT02636465
Title: Hypoxia in Flight Simulation in Obese Patients
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Deutsche Luft und Raumfahrt (Other Government)
Responsible Party: Sponsor
Other Study IDs: WI_105/2013
Record Dates: First submitted 2015-11-02; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Obesity, COPD, OHS
MeSH Terms: conditions — Obesity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- obese healthy adults: persons with BMI> 30 kg/m2
  Interventions: Other: flight simulationin obese healthy adults or obese patients with or without COPD, OHS
- obese COPD patients: COPD-patients (GOLD I-IV Group A-D) with BMI> 30 kg/m2
  Interventions: Other: flight simulationin obese healthy adults or obese patients with or without COPD, OHS
- OHS-patients: patients with defined OHS: BMI>30 kg/m2 and sleep related breathing disease, no COPD
  Interventions: Other: flight simulationin obese healthy adults or obese patients with or without COPD, OHS

INTERVENTIONS:
Other: flight simulationin obese healthy adults or obese patients with or without COPD, OHS
  Other Names: flight simulation

SUMMARY:
The purpose of this pilot study is to determine whether obese adults,obese (BMI>30 kg/m2) with obesity hypoventilation or obese COPD-patients do undergo oxygen desaturation under flight simulation and if the hypoxic altitude simulation test is as effective as the hypoxic chamber test.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* patients with COPD (GOLD I-IV Group A-D) with obesity (BMI> 30kg/m2), obese healthy adults with BMI> 30kg /m2, patients with Obesity hypoventilation syndrome
* informed consent provided

Exclusion Criteria:

* patients less than BMI <30 kg/m2 with or without COPD, OHS
* Age < 18 years
* pregnancy, lactation
* any medical, psychological or other condition restricting the patient's ability to provide informed consent
* participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese (BMI>30 kg/m2) healthy adults, obese patients with obesity hypoventilation Syndrome, obese patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
desaturation (SaO2 in %) in flight simulation in obese patients | one hour each patient

SECONDARY OUTCOMES:
desaturation (SaO2 in %) in hypoxic chamber test versus hypoxia altitude Simulation test | one hour each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Bethanien Hospital, Solingen, Germany

REFERENCES:
- [Background] Edvardsen A, Ryg M, Akero A, Christensen CC, Skjonsberg OH. COPD and air travel: does hypoxia-altitude simulation testing predict in-flight respiratory symptoms? Eur Respir J. 2013 Nov;42(5):1216-23. doi: 10.1183/09031936.00157112. Epub 2012 Dec 20. PMID 23258777
- [Background] Edvardsen A, Akero A, Christensen CC, Ryg M, Skjonsberg OH. Air travel and chronic obstructive pulmonary disease: a new algorithm for pre-flight evaluation. Thorax. 2012 Nov;67(11):964-9. doi: 10.1136/thoraxjnl-2012-201855. Epub 2012 Jul 5. PMID 22767877
- [Background] Edvardsen A, Akero A, Hardie JA, Ryg M, Eagan TM, Skjonsberg OH, Bakke PS. High prevalence of respiratory symptoms during air travel in patients with COPD. Respir Med. 2011 Jan;105(1):50-6. doi: 10.1016/j.rmed.2010.10.006. Epub 2010 Oct 25. PMID 20974527
- [Background] Howard LS. Last call for the flight simulation test? Eur Respir J. 2013 Nov;42(5):1175-7. doi: 10.1183/09031936.00037813. No abstract available. PMID 24178931
- [Background] Ahmedzai S, Balfour-Lynn IM, Bewick T, Buchdahl R, Coker RK, Cummin AR, Gradwell DP, Howard L, Innes JA, Johnson AO, Lim E, Lim WS, McKinlay KP, Partridge MR, Popplestone M, Pozniak A, Robson A, Shovlin CL, Shrikrishna D, Simonds A, Tait P, Thomas M; British Thoracic Society Standards of Care Committee. Managing passengers with stable respiratory disease planning air travel: British Thoracic Society recommendations. Thorax. 2011 Sep;66 Suppl 1:i1-30. doi: 10.1136/thoraxjnl-2011-200295. No abstract available. PMID 21856702